CLINICAL TRIAL: NCT01229098
Title: A Phase 2 Maximal Use Systemic Exposure Study Evaluating the Safety and Efficacy of Calcipotriol 50 mcg/g Plus Betamethasone 0.5 mg/g (as Dipropionate) Gel Applied Once Daily in Subjects With Extensive Psoriasis Vulgaris on the Scalp and Non-scalp Regions of the Body (Trunk and/or Limbs)
Brief Title: Effect of LEO 80185 Gel on the HPA Axis and Calcium Metabolism in Subjects With Extensive Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEO 80185-G24
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-03

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEO 80185 (Experimental)
  Interventions: Drug: LEO 80185 (Xamiol® gel/Taclonex® Scalp topical suspension)

INTERVENTIONS:
Drug: LEO 80185 (Xamiol® gel/Taclonex® Scalp topical suspension) — LEO 80185 (Taclonex® Scalp topical suspension/Xamiol® gel) Topical suspension applied once daily for up to 8 weeks

SUMMARY:
The purpose of this study is to evaluate the effect of once daily use of LEO 80185 gel on the hypothalamic-pituitary-adrenal (HPA) axis and calcium metabolism in subjects with extensive psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained following receipt of verbal and written information about the study prior to any trial related activities (including any wash-out period).
2. Age 18 years or above.
3. Either sex.
4. Any race or ethnicity.
5. Attending a hospital out-subject clinic or the private practice of a dermatologist for treatment of psoriasis vulgaris.
6. Clinical diagnosis of psoriasis vulgaris involving non scalp regions of the body (trunk and/or limbs) with or without involvement of the scalp.
7. At SV2 and Day 0 (Visit 1) a clinical diagnosis of psoriasis vulgaris which is:

   * amenable to topical treatment with a maximum of 100 g of study medication per week, and
   * of an extent of between 15 and 30% of the body surface area (BSA) excluding psoriasis on the face, genitals or skin folds.
   * a disease severity on the trunk and/or limbs graded as at least moderate according to the investigator's global assessment (IGA)
8. Subjects with normal HPA axis function at SV2 including a serum cortisol concentration above 5 mcg/dL before ACTH challenge test and above 18 mcg/dL 30 minutes after ACTH challenge test.
9. Albumin-corrected serum calcium, below the upper reference limit at SV2.
10. Females of child-bearing potential must have a negative urine pregnancy test result at baseline Visit SV2 and must agree to use a highly effective method of contraception during the study. Highly effective methods are defined as ones which results in a low failure rate (less than 1% per year) such as progestin-only formulations (implants, injectables), some intra-uterine devices, or vasectomised partner. Subjects must have used the contraceptive method continuously for at least 1 month prior to the pregnancy test and must continue using the contraceptive method for at least 1 week after the last application of study medication (or until study visit FU2 if applicable). A female is defined as not of child-bearing potential if she is postmenopausal (12 months with no menses without an alternative medical cause), or surgically sterile (tubal ligation/section, hysterectomy or bilateral ovariectomy).
11. Able to communicate with the investigator and understand and comply with the requirements of the study.

    Exclusion Criteria:
12. A history of serious allergy, allergic asthma or serious allergic skin rash
13. Known or suspected hypersensitivity to any medication (including ACTH/cosyntropin/tetracosactide) or to any component of the LEO 80185 gel or CORTROSYN.
14. Systemic treatment with corticosteroids (including inhaled and nasal steroids) within 12 weeks prior to SV2 and during the study.
15. Systemic treatment with biological therapies (marketed or not marketed), with a possible effect on psoriasis vulgaris within the following time period prior to Day 0 (Visit 1) and during the study:

    * etanercept - within 4 weeks prior to Visit 1
    * adalimumab, alefacept, infliximab -within 2 months prior to Visit 1
    * ustekinumab, briakinumab - within 4 months prior to Visit 1
    * experimental products - within 4 weeks/5 half-lives (whichever is longer) prior to Visit 1
16. Systemic treatment with therapies other than biologicals, with a possible effect on psoriasis vulgaris (e.g., retinoids, methotrexate, immunosuppressants) within 4 weeks prior to Visit 1 (Day 0) or during the study.
17. PUVA or Grenz ray therapy within 4 weeks prior to Visit 1 (Day 0) or during the study
18. UVB therapy within 2 weeks prior to Visit 1 (Day 0) or during the study.
19. Topical treatment with corticosteroids or vitamin D analogues (calcipotriol, calcitriol or tacalcitol) on any body location within 2 weeks prior to SV2 or during the study.
20. Any topical treatment of psoriasis vulgaris on the scalp or trunk and/or limbs (except for emollients and non-steroid medicated shampoos) within 2 weeks prior to Visit 1 (Day 0) or during the study.
21. Oral calcium supplements, vitamin D supplements, antacids, thiazide and/or loop diuretics, antiepileptics, diphosphonates or calcitonin within 4 weeks prior to SV2 and during the study. Note: Stable doses of oral vitamin D supplementation ≤400 IU/day is permitted provided there are no dose adjustments during the study period.
22. Planned initiation of, or changes to, concomitant medication that could affect psoriasis vulgaris (e.g., betablockers, antimalarials, lithium, ACE inhibitors) during the study.
23. Planned excessive exposure of treated areas to either natural or artificial sunlight (e.g. sunlamps etc.) during the study that may affect the psoriasis vulgaris.
24. Oestrogen therapy (including contraceptives) or any other medication known to affect cortisol levels or HPA axis integrity within 4 weeks prior to SV2 or during the study.
25. Cytochrome P450 3A4 (CYP 3A4) inducers (e.g., barbiturates, phenytoin, rifampicin) within 4 weeks prior to SV2 or during the study.
26. Systemic or topical cytochrome P450 3A4 (CYP 3A4) inhibitors (e.g., ketoconazole, itraconazole, metronidazole) within 4 weeks prior to SV2 or during the study. Topical ketoconazole within 2 weeks prior to SV2.
27. Hypoglycaemic sulfonamides within 4 weeks prior to the SV2 or during the study.
28. Antidepressant medications within 4 weeks prior to SV2 or during the study.
29. Not following nocturnal sleep patterns (e.g. night shift workers are excluded).
30. Known or suspected endocrine disorder that may affect the results of the ACTH challenge test.
31. Clinical signs or symptoms of Cushing's disease or Addison's disease.
32. Known or suspected diabetes mellitus.
33. Known or suspected cardiac disorders associated with abnormal QT intervals or rhythm disturbances including clinically significant bradycardia or tachycardia.
34. Known or suspected severe renal insufficiency or severe hepatic disorders.
35. Known or suspected disorders of calcium metabolism associated with hypercalcaemia.
36. Any clinically significant abnormality following review of screening laboratory tests (blood and spot urine samples), physical examination or blood pressure/heart rate measurement performed at SV2.
37. Current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis.
38. Any of the following conditions present on the study treatment areas: viral (e.g., herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, rosacea, acne vulgaris, acne rosacea, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, ulcers and wounds.
39. Other inflammatory skin diseases that may confound the evaluation of psoriasis vulgaris (e.g. seborrhoeic dermatitis, contact dermatitis and cutaneous mycosis).
40. Current participation in any other interventional clinical trial.
41. Previously enrolled in this trial (with the exception of subjects excluded due to hypocalcaemia prior to implementation of Consolidated Clinical Study Protocol 2).
42. Received any non-marketed drug substance (i.e., an agent which has not yet been made available for clinical use following registration) within 4 weeks or 5 half-lives (whichever is longer) prior to SV1.
43. Known or suspected of not being able to comply with the trial protocol (e.g., alcoholism, drug dependency or psychotic state).
44. Females who are pregnant, have a positive urine pregnancy test at baseline Visit SV2, or are breast-feeding. Females of child-bearing potential and wishing to become pregnant during the study or not using an adequate method of contraception during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Safety | Up to 8 weeks
  * Subjects with serum cortisol concentration of ≤18 mcg/dl at 30 minutes after ACTH-challenge [ Time Frame: Week 4 and week 8 ] [ Designated as safety issue: Yes ]
  * Change in albumin-corrected serum calcium from baseline [ Time Frame: Week 4 and week 8 ] [ Designated as safety issue: Yes ]
  * Change in 24-hour urinary calcium excretion from baseline [ Time Frame: Week 4 and week 8 ] [ Designated as safety issue: Yes ]
  * Change in urinary calcium:creatinine ratio from baseline [ Time Frame: Week 4 and week 8 ] [ Designated as safety issue: Yes ]

SECONDARY OUTCOMES:
Efficacy | Up to 8 weeks
  * Subjects with "Controlled disease" (i.e., "Clear" or "Almost clear") according to the investigator's global assessment of disease severity [ Time Frame: Weeks 2, 4, 8 ] [ Designated as safety issue: No ]
  * Pharmacokinetic parameters for calcipotriol, betamethasone dipropionate and any metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Shane Silver, MB, Principal Investigator — Dermadvances Research, 203 Edmonton Street, Winnipeg, Manitoba R3C 1R4 Canada
Locations (10):
- Canada (10):
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Dermadvances Research, Winnipeg, Manitoba
  - Alpha Clinical Research Centre, St. John's, Newfoundland and Labrador
  - Newlab Clinical Research, St. John's, Newfoundland and Labrador
  - Eastern Canada Cutaneous Research Associates Ltd., Halifax, Nova Scotia
  - Dermsearch, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - Institute of Cosmetic and Laser Surgery, Oakville, Ontario
  - Co-Medica Research Network Inc., Oshawa, Ontario
  - Oshawa Clinic, Oshawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silver S, Tuppal R, Gupta AK, Clonier F, Olesen M, Leeder R, Taraska V. Effect of calcipotriene plus betamethasone dipropionate topical suspension on the hypothalamic-pituitary-adrenal axis and calcium homeostasis in subjects with extensive psoriasis vulgaris: an open, non-controlled, 8-week trial. J Drugs Dermatol. 2013 Aug;12(8):882-7. PMID 23986161
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en